CLINICAL TRIAL: NCT06197399
Title: A Multicenter, Prospective, Randomized Controlled Trial Comparing the Efficacy of Detethering Surgery and Spinal Column Shortening Surgery in Adult Patients With Recurrent Tethered Cord Syndrome
Brief Title: A Randomized Controlled Trial for Surgical Treatment of Recurrent Adult Tethered Cord Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Chinese PLA General Hospital (Other); Seventh Medical Center of PLA Army General Hospital (Other); Chifeng Municipal Hospital (Other); The First Hospital of Hebei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XW-NS-RCT-RTCS
Record Dates: First submitted 2023-07-30; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Recurrent Adult Tethered Cord Syndrome
Keywords: Tethered cord syndrome; Detethering; Spinal Column Shortening
MeSH Terms: conditions — Neural Tube Defects

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Detethering Surgery (Experimental): Participants in this arm will undergo detethering surgery, a traditional surgical intervention that involves releasing the spinal cord from its abnormal attachment. All surgeries will be performed by trained and experienced neurosurgeons following standardized protocols.
  Interventions: Procedure: Detethering Surgery
- Spinal Column Shortening Surgery (Experimental): Participants in this arm will undergo spinal column shortening surgery, a surgical technique aimed at reducing tension on the spinal cord by shortening the vertebral column. All surgeries will be conducted by trained and experienced neurosurgeons following standardized protocols. Postoperative care will be similar in both arms to minimize confounding variables.
  Interventions: Procedure: Spinal Column Shortening Surgery

INTERVENTIONS:
Procedure: Detethering Surgery — Detethering surgery, or cord untethering, is a conventional surgical approach for treating tethered cord syndrome (TCS). It involves releasing the spinal cord from its abnormal attachment. During the surgical procedure, once the tethered area is identified, careful microsurgical techniques are used to separate the spinal cord from the surrounding abnormal tissue. This operation aims to alleviate the symptoms of TCS by removing the cause of tension on the spinal cord.
  Arms: Detethering Surgery
Procedure: Spinal Column Shortening Surgery — Spinal column shortening surgery is an innovative surgical approach that involves reducing the tension on the spinal cord by shortening the spinal column, effectively "untethering" the spinal cord indirectly. The procedure primarily involves the thoracolumbar region.The choice of this region for intervention offers several advantages: it is a safe distance from the previous detethering surgery area; it is closer to the conus medullaris of the spinal cord, ensuring better treatment effectiveness; and the impact on spinal mobility is minimal after internal fixation at this region. This technique is designed to alleviate TCS symptoms while minimizing the risk of postoperative cerebrospinal fluid (CSF) leakage, which is a common complication in direct untethering procedures for recurrent cases. All procedures will be conducted by trained and experienced neurosurgeons following standardized protocols.
  Arms: Spinal Column Shortening Surgery

SUMMARY:
This trial compares detethering surgery and spinal column shortening surgery, two treatments for adults with recurrent tethered cord syndrome (TCS), a neurological disorder where the spinal cord becomes abnormally attached to tissue. Detethering surgery carries a higher risk of postoperative complications such as cerebrospinal fluid (CSF) leakage, while spinal column shortening surgery's comparative efficacy is unclear. This study aims to clarify the optimal surgical management for recurrent TCS in adults, assessing postoperative complication rate and improvement of symptoms.

DETAILED DESCRIPTION:
This study is a multicenter, prospective, randomized controlled trial designed to compare the effectiveness and safety of detethering surgery and spinal column shortening surgery in adults diagnosed with recurrent tethered cord syndrome. TCS is a condition that causes neurological symptoms due to an abnormal attachment of the spinal cord to the surrounding tissue. The recurrent form in adults presents unique clinical challenges and limited treatment options.

Detethering surgery, a conventional treatment method, involves releasing the spinal cord from its abnormal attachment. While this technique directly addresses the cause of the condition, it also carries a high risk of cerebrospinal fluid (CSF) leakage, a severe postoperative complication.

Spinal column shortening surgery is a relatively new technique that aims to reduce tension on the spinal cord by shortening the vertebral column. It has been reported to offer a lower risk of CSF leakage, but its comparative efficacy to detethering surgery remains unclear due to limited evidence.

The proposed multicenter, prospective, randomized controlled trial aims to fill this knowledge gap by comparing the efficacy and safety of detethering surgery versus spinal column shortening surgery in adults with recurrent TCS. The results of this study will provide valuable insights into the optimal surgical management of adult patients with recurrent TCS, potentially improving patient outcomes, enhancing clinical practice, and guiding future research in this field.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have previously detethering surgery for primary tethered cord syndrome, including filum terminale untethering, dermoid or lipoma resection, with a recurrence of spinal cord tethering postoperatively.
* The presence of related clinical symptoms, including bowel and bladder dysfunction, sensory impairment, numbness, pain in the lower limbs, perineal or buttock area, motor dysfunction of the lower limbs, muscle weakness, and sexual dysfunction.
* Primary diagnosis of a thickened filum terminale, low-lying conus medullaris, meningocele, lipoma, dermoid, or spina bifida.

Exclusion Criteria:

* Patients with severe scoliosis at the thoracolumbar junction.
* Patients with severe osteoporosis or other conditions that contraindicate internal fixation.
* Patients with severe pressure ulcers or skin breakdown in the lumbar or thoracic region.
* Patients with severe systemic diseases that cannot tolerate surgery.
* Other cases deemed unsuitable for inclusion following evaluation by professional neurosurgeons.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of cerebrospinal fluid leakage | 7 days
  Postoperative Incidence of cerebrospinal fluid leakage

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) | 3 months, 6 months
  Postoperative lumbar and lower extremities VAS
12-item Short Form Health Survey (SF-12) | 3 months, 6 months
  Postoperative SF-12 evaluation
Muscle strength | 3 months, 6 months
  muscle strength of the lower extremities
Uroflow rate | 6 months
  Urodynamic test
Urodynamic test | 6 months
  Cystometry
Residual urine | 6 months
  Urodynamic test

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang C, Chang CC, Mummaneni PV, Yuan C, Dhall S, Jian F, Gupta N, Chou D. Spinal column shortening versus revision detethering for recurrent adult tethered cord syndrome: a preliminary comparison of perioperative and clinical outcomes. J Neurosurg Spine. 2020 Feb 7;32(6):958-964. doi: 10.3171/2019.12.SPINE19659. Print 2020 Jun 1. PMID 32032960
- [Background] Aldave G, Hansen D, Hwang SW, Moreno A, Briceno V, Jea A. Spinal column shortening for tethered cord syndrome associated with myelomeningocele, lumbosacral lipoma, and lipomyelomeningocele in children and young adults. J Neurosurg Pediatr. 2017 Jun;19(6):703-710. doi: 10.3171/2017.1.PEDS16533. Epub 2017 Mar 31. PMID 28362188
- [Background] Hsieh PC, Stapleton CJ, Moldavskiy P, Koski TR, Ondra SL, Gokaslan ZL, Kuntz C. Posterior vertebral column subtraction osteotomy for the treatment of tethered cord syndrome: review of the literature and clinical outcomes of all cases reported to date. Neurosurg Focus. 2010 Jul;29(1):E6. doi: 10.3171/2010.4.FOCUS1070. PMID 20594004
- [Background] McVeigh LG, Anokwute MC, Chen S, Jea A. Spinal column shortening for tethered cord syndrome: a systematic review and individual patient data meta-analysis. J Neurosurg Pediatr. 2022 Mar 4;29(6):624-633. doi: 10.3171/2022.1.PEDS21503. Print 2022 Jun 1. PMID 35245903
- [Background] O'Connor KP, Smitherman AD, Milton CK, Palejwala AH, Lu VM, Johnston SE, Homburg H, Zhao D, Martin MD. Surgical Treatment of Tethered Cord Syndrome in Adults: A Systematic Review and Meta-Analysis. World Neurosurg. 2020 May;137:e221-e241. doi: 10.1016/j.wneu.2020.01.131. Epub 2020 Jan 28. PMID 32001403